CLINICAL TRIAL: NCT03758092
Title: Cardiovascular Screening in 2-year Old Infants Born Small for Gestational Age Compared With Infants Born Adequate for Gestational Age
Brief Title: Cardiovascular Screening in Infants Born Small for Gestational Age
Acronym: CardioSGA
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Prof, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE 106/18
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Abnormalities; Small-for-gestational Age
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SGA vs AGA infants: infants, born at term (37+0/41+3 week gestation), aged 24 months, with a birth weight <10th percentile or between 10th and 90th percentile for sex, gestational age, and birth order, according to Italian neonatal anthropometric charts

SUMMARY:
Aims of this study were 1) to evaluate early CV abnormalities in infants born small for gestational age (SGA) at 24 months of age compared with age and sex-matched subjects that were born adequate for gestational age (AGA) 2) to investigate the effect of catch-up growth and the role of breastfeeding on CV risk.

DETAILED DESCRIPTION:
We consecutively enrolled 20 SGA infants, born at term (37+0/41+3 week gestation), aged 24 months, and 20 AGA, age- and sex-matched controls. SGA was defined as a birth weight <10th percentile for sex, gestational age and birth order, and AGA as a birth weight between the 10th and the 90th percentile, according to Italian neonatal anthropometric charts.

Clinical and anthropometric variables The infants' prenatal and neonatal data were retrospectively recorded, namely a history of gestational diabetes and hypertension, the presence of intrauterine growth restriction, maternal weight gain during pregnancy, Apgar score, gestational age and birth weight, length, and head circumference. All subjects' parents completed a questionnaire including family history, maternal smoking during pregnancy, breastfeeding duration. At the time of enrollment (24 months), anthropometric data were evaluated by trained physicians according to standard procedures and based on the WHO growth charts. Height, weight, systolic (SBP) and diastolic (DBP) blood pressure were measured. Body mass index (BMI) was calculated as weight (kg)/height(cm)2 and weight gain in the first 2 years of life was calculated as the delta between birth weight and weight at 24 months.

Echocardiographic assessment Transthoracic echocardiogram using a Vivid 7 Pro ultrasound scanner (General Electric Healthcare, USA) was performed by an expert pediatric cardiologist, blinded to patients' clinical data. Measurements of left ventricle (LV end-diastolic diameter, LVEDD; LV end-systolic diameter, LVESD; interventricular septum at end diastole, IVSD; LV posterior wall at end diastole, LVPWD), relative wall thickness (RWT), left atrium diameter (LAD), the maximum LA volume, LV ejection fraction, and tricuspid annular plane systolic excursion (TAPSE) were obtained according to established standards. LV mass (LVM) was derived from the Devereux formula and indexed to body surface area (left ventricular mass index, LVMI). Left ventricular output (LVO) was obtained with the velocity time integral (VTI) from a 5-chamber view and calculated as follows LVO=[(VTI)x(heart rate)x(cross-sectional area)] and indexed to body weight.

Using pulsed wave Doppler, mitral inflow velocities, peak early diastolic velocity (E), peak late diastolic velocity (A), and E/A ratio, were measured. Pulsed wave tissue Doppler of the lateral mitral annulus was used for the measurement of early peak diastolic mitral annular velocity (E'). The E/E' ratio was calculated. End-diastolic pressure (EDP) was calculated from the E/E' ratio with the formula EDP=1.91+1.24xE/E' (14) and the pressure-volume curve during diastole with the formula EDP = αxEDVβ (end-diastolic volume, EDV). Volume parameters were corrected to fixed values of EDP (V30 mmHg). The coefficient "β" (Beta), indicating the slope of the end-diastolic pressure-volume relationship (EDPVR), was calculated with the formula β=[Log10(EDP/30)]/[Log10(EDV/V30mmHg)].

Vascular assessment Vascular measurements were performed with a high-resolution ultrasonography (Esaote MyLab25TM Gold, Esaote, Italy) using a 8 mHz linear transducer and a 5 mHz convex transducer for the abdominal aorta, by an expert vascular surgeon blinded to patients' clinical status. CIMT, abdominal aortic diameter at maximum systolic expansion (Ds) and minimum diastolic expansion (Dd), brachial artery diameters, brachial artery peak systolic velocity (PSV) and end diastolic velocity (EDV) were measured as previously described and aortic strain (S), pressure strain elastic modulus (Ep), pressure strain normalized by diastolic pressure (Ep*) and brachial artery flow-mediated dilation (FMD) were calculated. While S is the mean strain of the aortic wall, Ep and Ep* are the mean stiffness (16). Arterial wall stiffness index (β index) was calculated with the formula: β index=ln(SBP/DBP)/[(Ds-Dd) /Dd)] (17) and systemic vascular resistance (dynes/s/cm2) with the formula: SVR=(mean BP- right atrial pressure)/LVO, with an estimated right atrial pressure of 5 mmHg. The brachial artery maximum diameter recorded following reactive hyperemia was reported as a percentage change of resting diameter (FMD = peak diameter - baseline diameter/baseline diameter).

ELIGIBILITY:
Inclusion Criteria:

* infants, 24-month old, born at term SGA or AGA

Exclusion Criteria:

* heart, respiratory, liver and kidney diseases, congenital malformations, genetic diseases, neonatal asphyxia, parenteral nutrition, congenital inborn errors of metabolism, and preterm and twin birth.

Ages: 24 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We consecutively enrolled 20 SGA infants, born at term (37+0-41+3 weeks gestation), aged 24 months, and 20 AGA, age- and sex-matched controls. SGA was defined as a birth weight <10th percentile for sex, gestational age and birth order, and AGA as a birth weight between the 10th and the 90th percentile, according to Italian neonatal anthropometric charts
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular structure | 24 months
  Heart structure
Cardiovascular function | 24 months
  Heart function

SECONDARY OUTCOMES:
catch-up growth | 24 months
  delta between body weight at 24 months and birth weight
breastfeeding duration | 24 months
  breastfeeding duration

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Maggiore della Carità - Clinica Pediatrica - Ambulatorio di Auxologia ed Endocrinologia Pediatrica, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker DJ, Osmond C, Golding J, Kuh D, Wadsworth ME. Growth in utero, blood pressure in childhood and adult life, and mortality from cardiovascular disease. BMJ. 1989 Mar 4;298(6673):564-7. doi: 10.1136/bmj.298.6673.564. PMID 2495113
- [Background] Ong KK, Ahmed ML, Emmett PM, Preece MA, Dunger DB. Association between postnatal catch-up growth and obesity in childhood: prospective cohort study. BMJ. 2000 Apr 8;320(7240):967-71. doi: 10.1136/bmj.320.7240.967. PMID 10753147
- [Background] Faienza MF, Brunetti G, Delvecchio M, Zito A, De Palma F, Cortese F, Nitti A, Massari E, Gesualdo M, Ricci G, Carbonara S, Giordano P, Cavallo L, Scicchitano P, Ciccone MM. Vascular Function and Myocardial Performance Indices in Children Born Small for Gestational Age. Circ J. 2016;80(4):958-63. doi: 10.1253/circj.CJ-15-1038. Epub 2016 Feb 10. PMID 26861187
- [Background] Iruretagoyena JI, Gonzalez-Tendero A, Garcia-Canadilla P, Amat-Roldan I, Torre I, Nadal A, Crispi F, Gratacos E. Cardiac dysfunction is associated with altered sarcomere ultrastructure in intrauterine growth restriction. Am J Obstet Gynecol. 2014 Jun;210(6):550.e1-7. doi: 10.1016/j.ajog.2014.01.023. Epub 2014 Jan 16. PMID 24440565
- [Background] Crispi F, Bijnens B, Figueras F, Bartrons J, Eixarch E, Le Noble F, Ahmed A, Gratacos E. Fetal growth restriction results in remodeled and less efficient hearts in children. Circulation. 2010 Jun 8;121(22):2427-36. doi: 10.1161/CIRCULATIONAHA.110.937995. Epub 2010 May 24. PMID 20497977
- [Background] Dratva J, Breton CV, Hodis HN, Mack WJ, Salam MT, Zemp E, Gilliland F, Kuenzli N, Avol E. Birth weight and carotid artery intima-media thickness. J Pediatr. 2013 May;162(5):906-11.e1-2. doi: 10.1016/j.jpeds.2012.10.060. Epub 2012 Dec 20. PMID 23260106